CLINICAL TRIAL: NCT05990790
Title: The Effect of Desflurane Versus Sevoflurane Versus Propofol on Postoperative Delirium in Elderly Patients Undergoing Moderate- to High-risk Major Noncardiac Surgery - a Prospective, Observer-blinded, Randomized, Clinical Trial
Brief Title: The Effect of Desflurane Versus Sevoflurane Versus Propofol on Postoperative Delirium
Acronym: RAPID-II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAPIDII_01
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Delirium; Major Noncardiac Surgery; Postoperative Cognitive Dysfunction
Keywords: Propofol; Sevoflurane; Desflurane
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Desflurane; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Desflurane Group (Experimental): After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of desflurane with an intraoperative goal of bispectral index (BIS) 50±10.
  Interventions: Drug: Desflurane
- Sevoflurane Group (Active Comparator): After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of sevoflurane with an intraoperative goal of bispectral index (BIS) 50±10.
  Interventions: Drug: Sevoflurane
- Propofol Group (Active Comparator): After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of propofol with an intraoperative goal of bispectral index (BIS) 50±10.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of desflurane with an intraoperative goal of bispectral index (BIS) 50±10.
  Arms: Desflurane Group
Drug: Sevoflurane — After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of sevoflurane with an intraoperative goal of bispectral index (BIS) 50±10.
  Arms: Sevoflurane Group
Drug: Propofol — After induction of anesthesia, maintenance of anesthesia will be performed using goal-directed administration of propofol with an intraoperative goal of bispectral index (BIS) 50±10.
  Arms: Propofol Group

SUMMARY:
Patients over the age of 65 years are at increased risk for developing delirium after noncardiac surgeries, resulting in increased morbidity and mortality. The prevention of postoperative delirium has been classified as a public health priority. However, so far data regarding possible intraoperative interventions to reduce the incidence of postoperative delirium is very scarce. Due to the more rapid wash-in and wash-out times of desflurane as compared to sevoflurane or propofol it seems reasonable that desflurane might be beneficial for the prevention of postoperative delirium. Therefore, we evaluate the effect of maintenance of anesthesia using desflurane, sevoflurane or propofol on postoperative delirium in elderly patients undergoing moderate- to high-risk major noncardiac surgery.

DETAILED DESCRIPTION:
Background: Postoperative delirium occurs in approximately 25% of patients over the age of 60 years undergoing major noncardiac surgery and is significantly associated with an increase in postoperative neurocognitive decline, morbidity, and mortality. The prevention of postoperative delirium has been classified as a public health priority. However, so far data regarding possible intraoperative interventions to reduce the incidence of postoperative delirium is very scarce. Previous small studies compared the effect of administration of sevoflurane versus propofol for maintenance of anesthesia on postoperative delirium and found beneficial effects of volatile anesthesia for the prevention of postoperative delirium. Furthermore, in small studies the administration of desflurane led to significantly shorter recovery periods after noncardiac surgery as compared to sevoflurane. Due to the more rapid wash-in and wash-out times of desflurane as compared to sevoflurane or propofol it seems reasonable that desflurane might be beneficial for the prevention of postoperative delirium. Therefore, we evaluate the effect of maintenance of anesthesia using desflurane, sevoflurane or propofol on postoperative delirium in elderly patients undergoing moderate- to high-risk major noncardiac surgery.

Methods: We will include 1332 patients ≥ 65 years of age undergoing moderate- to high-risk major noncardiac surgery lasting at least two hours in this prospective observer-blinded randomized controlled clinical trial. After induction of anesthesia patients will be randomly assigned to receive desflurane, sevoflurane or propofol for maintenance of anesthesia. Our primary outcome will be the incidence of postoperative delirium in the first five postoperative days. Postoperative delirium will be diagnosed using the 3D-CAM or 3D-CAM-ICU in the morning and evening of the first five postoperative days as appropriate assessed by blinded study personnel. Two-interim analyses after 1/3 and 2/3 of recruitment are pre-planned.

Statistics: The primary outcome, the incidence of postoperative delirium in the first five postoperative days, will be compared between the groups using a Chi-Square-test as well as a logistic regression model for the incidence of postoperative delirium will be performed accounting for randomized group, age and other possible confounding factors.

Level of originality: Data regarding possible intraoperative interventions for the prevention of postoperative delirium are scarce. In detail, the effects of commonly used anesthetics on the incidence of postoperative delirium and neurocognitive dysfunction have only been studied in retrospective analyses or small prospective studies, which showed inconsistent results. Nevertheless, delirium is a major event after surgery and is associated with postoperative complications, worse neurocognitive recovery and increased mortality, especially in elderly patients. Thus, the results of this trial will help to choose the right anesthetic according to individual patients' requirements to reduce the risk for postoperative delirium in future.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* ≥65 years of age
* Scheduled for elective major noncardiac surgery with estimated time of surgery ≥ 2 hours

Exclusion Criteria:

* Patients undergoing emergency surgery
* BMI > 45 kg/m^2
* History of diagnosed dementia
* Language, vision, or hearing impairments that may compromise cognitive assessments
* History of malignant hyperthermia
* History of structural muscle disease
* History of organ transplantation (kidney, liver, lung, heart)
* Patients undergoing hyperthermic intraperitoneal chemotherapy
* ICU patients undergoing surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1332 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | First five postoperative days
  Delirium will be assessed via 3D-cognitive assessment method (3D-CAM) test as early in the morning as practical and in the early evening for the initial five postoperative days while the patients remain hospitalized according to current recommendations. In patients in the intensive care unit (ICU), we will perform the 3D-CAM-ICU. Any positive CAM test will be considered evidence of delirium, which will be analyzed dichotomously.

SECONDARY OUTCOMES:
Digit Symbol-Substitution-Test for the incidence of postoperative cognitive dysfunction (POCD) | First five postoperative days
  POCD will be assessed using the Digit-Symbol-Substitution-Test (DSST). The occurrence of POCD will be defined when a patient has a Z score on two or all tests or the combined Z score is below -1.96 standard deviation (SD).
Trail Making Test (TMT) for the incidence of postoperative cognitive dysfunction (POCD) | First five postoperative days
  POCD will be assessed using the Trail Making Test (TMT). The occurrence of POCD will be defined when a patient has a Z score on two or all tests or the combined Z score is below -1.96 standard deviation (SD).
Postoperative need of supplemental oxygen | During PACU/ICU stay after surgery (max. of first 24 hours after surgery)
  We will record postoperative need for administration of supplemental oxygen to maintain a SpO2 of 93% during PACU or ICU stay.
Length of stay in ICU | First 30 days after surgery
  Length of stay in ICU after surgery.
Incidence of Postoperative nausea and vomiting in the early postoperative period | First two hours after surgery
  Episode of nausea and/or vomiting within the first two hours after surgery
Incidence of Postoperative nausea and vomiting in the late postoperative period | First five postoperative days
  Episode of nausea and/or vomiting from two hours after surgery until the fifth postoperative day.
Intraoperative hypotension | During surgery
  Intraoperative duration of mean arterial pressure <65mmHg and overall amount of intraoperatively administered catecholamines (including phenylephrine, norepinephrine, epinephrine, etilefrine, ephedrine).
Death within 5 days after surgery | First five postoperative days
  Mortality in the first five postoperative days.

OTHER OUTCOMES:
Days at home in the first month after surgery | First 30 days after surgery
  Number of days at home within the first 30 postoperative days.
Long-term postoperative cognitive dysfunction | One year after surgery
  Long-term postoperative cognitive dysfunction will be assessed via Montreal cognitive assessment (MoCA). We will assess the baseline MoCA a day before surgery and one year after surgery via phone interview. Minimum score of the MoCA is 0 points. Maximum score of the MoCA is 22 points. Postoperative cognitive dysfunction is defined as a reduction of at least 2 points as compared to baseline.
Postoperative IL-6 concentrations (pg/ml) | First two postoperative days
  Postoperative area under the curve (AUC) within the first two postoperative days of concentrations of Interleukin 6 (IL-6).
Postoperative PCT concentrations (ng/ml) | First two postoperative days
  Postoperative area under the curve (AUC) within the first two postoperative days of concentrations of Procalcitonin (PCT).
Postoperative CRP concentrations (mg/dl) | First two postoperative days
  Postoperative area under the curve (AUC) within the first two postoperative days of concentrations of C-reactive protein (CRP).
Postoperative Copeptin concentrations (pmol/L) | First two postoperative days
  AUC within the first two postoperative days of concentrations of Copeptin.
Postoperative TnT concentrations (ng/L) | First two postoperative days
  AUC within the first two postoperative days of concentrations of TnT.
Postoperative NT-proBNP concentrations (pg/ml) | First two postoperative days
  AUC within the first two postoperative days of concentrations of NT-proBNP.
Postoperative S100-B concentrations (µg/L) | First two postoperative days
  AUC within the first two postoperative days of concentrations of S100-B.
Postoperative NSE concentrations (µg/L) | First two postoperative days
  AUC within the first two postoperative days of concentrations of NSE.
All-cause death within one year after surgery | One year after surgery
  All cause one-year mortality.
Sub-Study Advanced Neurobiomarkers | Baseline and third postoperative day.
  Difference of serum Neurofilament light-chain (sNFL)and Glial fibrillary acidic protein (GFAP) concentrations between the groups.
Sub-Study Analgesia Nociception Index (ANI) | Intraoperative
  Association between ANI and postoperative delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Reiterer, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taschner A, Fleischmann E, Kabon B, Sinner B, Eckhardt C, Horvath K, Adamowitsch N, Hantakova N, Hochreiter B, Zotti O, Fraunschiel M, Graf A, Reiterer C; RAPID II Trial investigators. Effect of desflurane, sevoflurane or propofol on the incidence of postoperative delirium in older adults undergoing moderate- to high-risk major non-cardiac surgery: study protocol for a prospective, randomised, observer-blinded, clinical trial (RAPID-II trial). BMJ Open. 2024 Nov 27;14(11):e092611. doi: 10.1136/bmjopen-2024-092611. PMID 39609026